CLINICAL TRIAL: NCT00921505
Title: The Effect of Ibuprofen, Paracetamol and Their Combination on Reactive Oxygen Species (ROS)- Production in Leukocytes and Platelet Activation
Brief Title: Effect of Ibuprofen, Paracetamol and Their Combination on Radical Oxygen Species (ROS) Production
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ullevaal University Hospital (Other)
Collaborators: University of Oslo (Other)
Responsible Party: Professor Torstein Lyberg, Ullevaal University Hospital
Organization: Oslo University Hospital (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: PARIBU-024; EudraCT No. 2009-009036-77
Record Dates: First submitted 2009-06-15; First posted 2009-06-16 (Estimated); Last update posted 2011-07-06 (Estimated); Status verified 2009-03

CONDITIONS: Pain
Keywords: Acetaminophen; Ibuprofen; Platelets; Leukocytes; Oxygen species; Humans; Blood Platelets; Reactive Oxygen Species; Platelet Activation
MeSH Terms: conditions — Pain | interventions — Ibuprofen; Acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Ibuprofen 400 mg (Active Comparator): Ibuprofen oral single dose
  Interventions: Drug: Ibuprofen
- Ibuprofen 1200 mg (Active Comparator): Ibuprofen oral single dose
  Interventions: Drug: Ibuprofen
- Paracetamol (acetaminophen) 1000 mg (Active Comparator): Paracetamol (acetaminophen) oral single dose
  Interventions: Drug: Paracetamol (acetaminophen) 1000 mg
- Ibuprofen 400 mg + paracetamol 1000 mg (Active Comparator): Paracetamol (acetaminophen) + ibuprofen oral single dose
  Interventions: Drug: Paracetamol + ibuprofen

INTERVENTIONS:
Drug: Ibuprofen — Tablet ibuprofen 400 mg oral single dose (1 tablet)
  Other Names: Ibumetin; ATC code: M01A E01
  Arms: Ibuprofen 400 mg
Drug: Ibuprofen — Tablets (2 x 600 mg) oral single dose (2 tablets)
  Other Names: Ibumetin; ATC code: M01A E01
  Arms: Ibuprofen 1200 mg
Drug: Paracetamol (acetaminophen) 1000 mg — Tablets (2 x 500 mg) oral single dose (2 tablets)
  Other Names: Paracetamol; Acetaminophen; ATC code: N02B E01
  Arms: Paracetamol (acetaminophen) 1000 mg
Drug: Paracetamol + ibuprofen — Tablets (ibuprofen 400 mg + paracetamol (acetaminophen) 2 x 500 mg) single oral dose (3 tablets)
  Other Names: Ibumetin; Ibuprofen; ATC code: M01A E01; Paracetamol; Acetaminophen; ATC code: N02B E01
  Arms: Ibuprofen 400 mg + paracetamol 1000 mg

SUMMARY:
The purpose of this study is to determine whether paracetamol, ibuprofen or their combination can modify generation of radical oxygen species (ROS) from stimulated neutrophils.

DETAILED DESCRIPTION:
Non-steroidal anti-inflammatory drugs (NSAID) are used to alleviate clinical inflammatory symptoms (e.g. pain, swelling and reduced function). Leukocytes, upon activation during inflammatory states, generate radical oxygen species (ROS) which primarily are intended for host defence against invading pathogens. Certain NSAID can modify the generation of ROS from stimulated neutrophils ranging form increased production to reduced production. Preliminary experiments in our laboratory have shown that different NSAIDs have opposing effects on the ability of leukocytes (granulocytes and monocytes) to produce ROS upon a standardized stimulus, i.e. phorbol myristate acetate (PMA). Paracetamol has a marked inhibitory effect and ibuprofen has a facilitating effect on ROS production. An inhibitory effect of paracetamol was also seen when examining platelet activation markers, whereas acetylsalicylic acid showed a clear enhancing effect in this respect. We want to examine if intake of paracetamol or ibuprofen in vivo have similar effects on leukocyte ROS production and platelet activation, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers of both sexes (ASA type I).
* Females who are not pregnant or plan conception. (A pregnancy test will be conducted before each test day)
* Persons who have not used analgesics for 3 days prior to the blood sampling.
* Persons without known active peptic ulcer or gastrointestinal bleeding.
* Persons without any known hypersensitivity for NSAIDs.
* Persons under no other drug treatment than contraceptives.
* Age 18 to 35 years of Caucasian origin

Exclusion Criteria:

* Pregnancy during the test period.
* Development of active peptic ulcer during the test period.
* Change in medication status during the test period (after inclusion).

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 7 (Estimated)
Dates: Start 2009-05; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Leukocyte radical oxygen species (ROS) production | 24 hours for each crossover event

SECONDARY OUTCOMES:
Platelet activation status | 24 hours for each crossover event

CONTACTS AND LOCATIONS:
Overall Officials: Torstein Lyberg, DDS, MD, Study Director — Ullevaal University Hospital
Locations (1):
- Ullevaal University Hospital, Oslo, Norway

REFERENCES:
- [Background] Stritesky Larssen K, Lyberg T. Oxidative status--age- and circadian variations?--a study in leukocytes/plasma. Neuro Endocrinol Lett. 2006 Aug;27(4):445-52. PMID 16891997
- [Background] Nagata M. Inflammatory cells and oxygen radicals. Curr Drug Targets Inflamm Allergy. 2005 Aug;4(4):503-4. doi: 10.2174/1568010054526322. PMID 16101529
- [Background] Nielsen VG, Webster RO. Inhibition of human polymorphonuclear leukocyte functions by ibuprofen. Immunopharmacology. 1987 Feb;13(1):61-71. doi: 10.1016/0162-3109(87)90027-0. PMID 3032852